CLINICAL TRIAL: NCT06408415
Title: A Study of the Higher Cognitive Functions of the Human Brain Based on the Use of Hyperflexible Neural Electrode-cortex for Single-neuron Activity Recording
Brief Title: A Study of the Higher Cognitive Functions of the Human Brain With Single-neuron Activity Recording
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Xuehai Wu, Professor, Huashan Hospital, Huashan Hospital
Other Study IDs: KY2024-638
Record Dates: First submitted 2024-04-26; First posted 2024-05-10 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Cognition
Keywords: Electrodes, Implanted; higher cognitive function; single neural activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study aims to investigate that neural activity of higher cognitve function of human brain with hyperflexible neural electrode-cortex

DETAILED DESCRIPTION:
In this study, patients who need intracerebral puncture and indwelling drainage tube, such as intracerebral hemorrhage and hydrocephalus, will be recruited. Before implanting electrodes, patients will be trained to do higher cognitive function tasks.During operation, electrode will be implanted accompanied by placing drainage tube. After operation, patients will perform tasks, while electrophysiological signals will be collected. At the end of study, electrode will be removed.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-70 years old.
2. have selective or confine operation indications:spontaneous basal ganglia hemorrhage or lobar hemorrhage that need catheter aspiration and drainage;hydrocephalus that need V-P shunt; need placing ommaya.
3. GCS score 12-15; must be able to communicate with investigators in Mandarin and comply with study requirements.
4. volunteered to participate in this study and sign informed consent.

Exclusion Criteria:

1. have severe cognitive dysfunction.
2. have psychiatric disorders, such as depression, anxiety disorders and schizophrenia.
3. long-term use of special medications, such as hormones, immunosuppressant, and anticoagulants.
4. be allergic to surgery instruments or medications.
5. have general anesthesia, surgery contraindications.
6. have acute cardiac infarction or heart arrest within 6 months.
7. have other neurosurgery contraindications assessed by investigators.
8. lactation or pregnancy.
9. have serious systemic disease or organ dysfunctions that affects study outcome or visits.
10. participate in other ongoing clinical trials.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients received treatments in Huashan hospital
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
recording local field potentiation | through study completion, an average of 2 year
  The mechanism of higher cognitive functions will be investigated by analysing characteristics of local field potentiation which is correlated with higher cognitive functions tasks, such as events related potential, information coding, etc.
recording single neural spikes | through study completion, an average of 2 year
  The mechanism of higher cognitive functions will be investigated by analysing characteristics of single neural spikes which is correlated with higher cognitive functions tasks, such as firing frequency, events related potential, information coding, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Xuehai Wu, Ph.D., Principal Investigator — Department of Neurosurgery, Huashan Hospital, Fudan University
Locations (1):
- Department of Neurosurgery, Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China